CLINICAL TRIAL: NCT06890533
Title: A Phase Ⅲ, Randomized, Double-Blind, Placebo- and Active-controlled Study of YZJ-4729 Tartrate Injection for the Treatment of Moderate to Severe Pain After Abdominal Surgery
Brief Title: A Study of YZJ-4729 Tartrate Injection for the Treatment of Pain After Abdominal Surgery
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Haiyan Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YZJ-4729-3-01
Record Dates: First submitted 2025-03-11; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental Group 1 (Experimental)
  Interventions: Drug: Experimental: YZJ-4729
- Experimental Group 2 (Experimental)
  Interventions: Drug: Experimental: YZJ-4729
- Placebo Comparator (Placebo Comparator)
  Interventions: Drug: Placebo Comparator: Saline
- Active Comparator (Active Comparator)
  Interventions: Drug: Active Comparator: Morphine

INTERVENTIONS:
Drug: Experimental: YZJ-4729 — Loading dose + demand dose
  Arms: Experimental Group 1; Experimental Group 2
Drug: Placebo Comparator: Saline — Loading dose + demand dose
  Arms: Placebo Comparator
Drug: Active Comparator: Morphine — Loading dose + demand dose
  Arms: Active Comparator

SUMMARY:
The primary objective is to evaluate the analgesic efficacy and safety of IV YZJ-4729 Tartrate Injection in patients with acute postoperative pain following abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to understand the study purpose and cooperate with the study procedures of this trial, voluntarily provide written informed consent
2. Body mass index (BMI) ≥18 kg/m2 and ≤28 kg/m2.
3. ASA I - II
4. Experiences a pain intensity rating of moderate to severe acute pain following abdominal surgery, with a pain intensity score of ≥4 on a Numeric Rating Scale (NRS) within 4 hours post-surgery

Exclusion Criteria:

1. Allergy to opioids and other medications that may be used during the trial.
2. Nervous system disorders (e.g. epilepsy)
3. Psychiatric disorders (e.g. depression)
4. History of difficult airways
5. Random blood glucose ≥11.1 mmol/L
6. Uncontrolled blood pressure [e.g., hypertension (systolic blood pressure ≥160 mmHg, diastolic blood pressure ≥100 mmHg)，or hypotension(systolic blood pressure <90 mmHg)]
7. Abnormal pulse oxygen saturation (SpO2 <90 %)
8. Abnormal liver function or renal function
9. Used agents that could affect the analgesic response
10. Used agents that could affect drug metabolism
11. Has previously participated in another YZJ-4729 clinical study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
the Sum of Pain Intensity Differences Over 24 Hours at rest | 24 hours
  Pain intensity will be evaluated using an 11-point (0-10) Numeric Pain Rating Scale (NRS), with higher numbers indicating a higher pain intensity, administered over 24 hours.

SECONDARY OUTCOMES:
The Time to first using rescue analgesics | 24 hours
The proportion of subjects using rescue analgesics | 24 hours
The number of times for rescue analgesics using | 24 hours
The cumulative dose used of rescue analgesics | 24 hours
the resting Sum of Pain Intensity Differences Over 6、12、18、12-24 Hours | 24 hours
the active Sum of Pain Intensity Differences Over 6、12、18、24、12-24 Hours | 24 hours
Participant satisfaction scores for analgesia treatment | 24 hours
  Participants recalled the postoperative analgesia effect and rated their satisfaction on a scale of 1 to 5, with 1 representing dissatisfied and 5 representing very satisfied.
Investigator satisfaction scores for analgesia treatment | 24 hours
  Postoperative analgesia was evaluated by investigators. The scale ranges from 1 to 5, with 1 being dissatisfied and 5 being very satisfied.

CONTACTS AND LOCATIONS:
Locations (49):
- China (49):
  - Cangzhou Central Hospital, Cangzhou
  - Cangzhou People's Hospital, Cangzhou
  - Changde First People's Hospital, Changde
  - Changsha Hospital Affiliated to Hunan University, Changsha
  - The Fourth Hospital OF Changsha, Changsha
  - The Third Xiangya Hospital of Central South University, Changsha
  - Sichuan Provincial People's Hospital, Chengdu
  - The Second People's Hospital of Chengdu, Chengdu
  - The Third People's Hospital of Chengdu, Chengdu
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing
  - The First Hospital of Jilin University, Ch’ang-ch’un
  - Affiliated Zhongshan Hospital of Dalian University, Dalian
  - Deyang People's Hospital, Deyang
  - Dongguan People's Hospital, Dongguan
  - Ganzhou People's Hospital, Ganzhou
  - The First People's Hospital of Guangyuan, Guangyuan
  - Guangdong Province Traditional Chinese Medical Hospital, Guangzhou
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou
  - The First Affiliated Hospital of Jinan University, Guangzhou
  - Haikou People's Hospital, Haikou
  - The Fourth Affiliated Hospital of Harbin Medical University, Ha’erbin
  - The Second People's Hospital of Hefei, Hefei
  - The First Affiliated Hospital of University of South China, Hengyang
  - Huzhou Central Hospital, Huzhou
  - The First Hospital of Jiaxing, Jiaxing
  - Liuzhou People's Hospital, Liuchow
  - Liuzhou Workers' Hospital, Liuchow
  - Luoyang Central Hospital, Luoyang
  - Ma'anshan People's Hospital, Ma’anshan
  - Mianyang Central Hospital, Mianyang
  - JiangXi Provincial People's Hospital, Nanchang
  - The Second Nanning People's Hospital, Nanning
  - The Second People's Hospital of Neijiang, Neijiang
  - Ningbo Medical Center Lihuili Hospital, Ningbo
  - Qingdao Central Hospital of Rehabilitation University, Qingdao
  - Shanghai First Maternity and Infant Hospital, Shanghai
  - Shanghai Fourth People's Hospital, Shanghai
  - Taizhou People's Hospital, Taizhou
  - The Second Hospital of Tianjin Medical University, Tianjin
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Wuhan Third Hospital, Wuhan
  - Affiliated Hospital of Jiangnan University, Wuxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - Zhongshan Hospital Xiamen University, Xiamen
  - The Second People's Hospital of Yibin, Yibin
  - Zhangzhou Municipal of Fujian Province, Zhangzhou
  - Henan Provincial People's Hospital, Zhengzhou
  - Zhuzhou Central Hospital, Zhuzhou